CLINICAL TRIAL: NCT03760146
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A 20-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN PNEUMOCOCCAL VACCINE-NAÏVE ADULTS 18 YEARS OF AGE AND OLDER
Brief Title: Trial to Evaluate the Safety and Immunogenicity of a 20-valent Pneumococcal Conjugate Vaccine in Pneumococcal Vaccine-naïve Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B7471007; 2018-004279-11 (EudraCT Number)
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Results first posted 2020-12-29 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 60 years and above 20vPnC/Saline (Experimental): 20vPnC and saline
  Interventions: Biological: 20vPnC; Other: Saline
- 60 years and above 13vPnC/PPSV23 (Active Comparator): 13vPnC and PPSV23
  Interventions: Biological: 13vPnC; Biological: PPSV23
- 50 through 59 years of age 20vPnC (Experimental): 20vPnC
  Interventions: Biological: 20vPnC
- 18 through 49 years of age 20vPnC (Experimental): 20vPnC
  Interventions: Biological: 20vPnC
- 50 through 59 years of age 13vPnC (Active Comparator): 13vPnC
  Interventions: Biological: 13vPnC
- 18 through 49 years of age 13vPnC (Active Comparator): 13vPnC
  Interventions: Biological: 13vPnC

INTERVENTIONS:
Biological: 20vPnC — 20vPnC
  Arms: 18 through 49 years of age 20vPnC; 50 through 59 years of age 20vPnC; 60 years and above 20vPnC/Saline
Biological: 13vPnC — Pneumococcal conjugate vaccine
  Arms: 18 through 49 years of age 13vPnC; 50 through 59 years of age 13vPnC; 60 years and above 13vPnC/PPSV23
Biological: PPSV23 — Pneumococcal polysaccharide vaccine
  Other Names: Pneumovax 23
  Arms: 60 years and above 13vPnC/PPSV23
Other: Saline — Placebo
  Arms: 60 years and above 20vPnC/Saline

SUMMARY:
A Phase 3, Randomized, Double-Blind Trial to Evaluate the Safety and Immunogenicity of a 20-valent Pneumococcal Conjugate Vaccine in Pneumococcal Vaccine-Naïve Adults

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults >/= 18 years of age (from the 18th birthday) at enrollment and older.
2. Adults determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study, including adults with preexisting stable disease, defined as disease not requiring significant change in therapy in the previous 6 weeks or hospitalization for worsening disease within 12 weeks before receipt of investigational product.
3. Negative urine pregnancy test at Visit1 for all subjects who are of childbearing potential.

Exclusion Criteria:

1. Previous vaccination with any licensed or investigational pneumococcal vaccine, or planned receipt through study participation.
2. History of microbiologically proven invasive disease caused by S pneumoniae.
3. Serious chronic disorder including metastatic malignancy, severe chronic obstructive pulmonary disease (COPD) requiring supplemental oxygen, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the subject from participating in the study.
4. Pregnant female subjects or breastfeeding female subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3902 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (66):
- United States (59):
  - Accel Research Sites, Birmingham, Alabama
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - East Valley Gastroenterology and Hepatology Associates, Chandler, Arizona
  - The Pain Center of Arizona, Peoria, Arizona
  - MedPharmics, LLC, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - Nature Coast Clinical Research, Crystal River, Florida
  - Accel Research Sites - Clinical Research Unit, DeLand, Florida
  - Research Centers of America, LLC, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Qps-Mra, Llc, South Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Meridian Clinical Research LLC, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Axtell Clinic, P.A., Newton, Kansas
  - Heartland Research Associates, LLC, Newton, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Northwest Family Physicians, Wichita, Kansas
  - Meridian Clinical Research, LLC, Rockville, Maryland
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Meridian Clinical Research LLC, Omaha, Nebraska
  - ActivMed Practices & Research, Inc., Portsmouth, New Hampshire
  - United Medical Associates, Binghamton, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - PharmQuest, Greensboro, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center (CCHMC), Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Omega Medical Research, Warwick, Rhode Island
  - Meridian Clinical Research, LLC, Dakota Dunes, South Dakota
  - Tekton Research, Inc., Austin, Texas
  - Bellaire Doctor's Clinic, Bellaire, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Benchmark Research, Fort Worth, Texas
  - HealthFirst Medical Group, Fort Worth, Texas
  - Ventavia Research Group, LLC, Keller, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Ventavia Research Group, LLC, Spring, Texas
  - DM Clinical Research, Tomball, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - J. Lewis Research Inc. / Foothill Family Clinic Draper, Draper, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc. - Jordan River Family Medicine, South Jordan, Utah
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington
- Sweden (7):
  - Ladulaas Kliniska Studier, Borås
  - Infektionskliniken Malarsjukhuset, Eskilstuna
  - ProbarE i Lund, Lund
  - Avdelningen för kliniska prövningar, Örebro
  - Karolinska Trial Alliance, KTA Prim, Stockholm
  - Akardo Med Site, Stockholm
  - Akademiska Sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Sabharwal C, Sundaraiyer V, Peng Y, Moyer L, Belanger TJ, Gessner BD, Jodar L, Jansen KU, Gruber WC, Scott DA, Watson W. Immunogenicity of a 20-valent pneumococcal conjugate vaccine in adults 18 to 64 years old with medical conditions and other factors that increase risk of pneumococcal disease. Hum Vaccin Immunother. 2022 Nov 30;18(6):2126253. doi: 10.1080/21645515.2022.2126253. Epub 2022 Nov 11. PMID 36368038
- [Derived] Essink B, Sabharwal C, Cannon K, Frenck R, Lal H, Xu X, Sundaraiyer V, Peng Y, Moyer L, Pride MW, Scully IL, Jansen KU, Gruber WC, Scott DA, Watson W. Pivotal Phase 3 Randomized Clinical Trial of the Safety, Tolerability, and Immunogenicity of 20-Valent Pneumococcal Conjugate Vaccine in Adults Aged >/=18 Years. Clin Infect Dis. 2022 Aug 31;75(3):390-398. doi: 10.1093/cid/ciab990. PMID 34940806
- [Derived] Mt-Isa S, Abderhalden LA, Musey L, Weiss T. Matching-adjusted indirect comparison of pneumococcal vaccines V114 and PCV20. Expert Rev Vaccines. 2022 Jan;21(1):115-123. doi: 10.1080/14760584.2021.1994858. Epub 2021 Oct 27. PMID 34672224
- [Derived] Perdrizet J, Santana CFS, Senna T, Alexandre RF, Sini de Almeida R, Spinardi J, Wasserman M. Cost-effectiveness analysis of replacing the 10-valent pneumococcal conjugate vaccine (PCV10) with the 13-valent pneumococcal conjugate vaccine (PCV13) in Brazil infants. Hum Vaccin Immunother. 2021 Apr 3;17(4):1162-1172. doi: 10.1080/21645515.2020.1809266. Epub 2020 Sep 23. PMID 32966176
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471007

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 20vPnC/Saline: Participants aged 60 years and above were randomized to receive a single dose of 0.5 milliliter (mL) intramuscular injection of 20-valent pneumococcal vaccine (20vPnC) at Vaccination 1 (Day 1) and a single dose of 0.5 mL intramuscular injection of saline at Vaccination 2 (28 to 42 days after Vaccination 1).
- Cohort 1: 13vPnC/PPSV23: Participants aged 60 years and above were randomized to receive a single dose of 0.5 mL intramuscular injection of 13-valent pneumococcal vaccine (13vPnC) at Vaccination 1 (Day 1) and a single dose of 0.5 mL intramuscular injection of 23-valent pneumococcal polysaccharide vaccine (PPSV23) at Vaccination 2 (28 to 42 days after vaccination 1).
- Cohort 2: 20vPnC: Participants aged 50 through 59 years were randomized to receive a single dose of 0.5 mL intramuscular injection of 20vPnC (Day 1).
- Cohort 2: 13vPnC: Participants aged 50 through 59 years were randomized to receive a single dose of 0.5 mL intramuscular injection of 13vPnC (Day 1).
- Cohort 3: 20vPnC: Participants aged 18 through 49 years were randomized to receive a single dose of 0.5 mL intramuscular injection of 20vPnC (Day 1).
- Cohort 3: 13vPnC: Participants aged 18 through 49 years were randomized to receive a single dose of 0.5 mL intramuscular injection of 13vPnC (Day 1).
Period: Overall Study
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23 | Cohort 2: 20vPnC | Cohort 2: 13vPnC | Cohort 3: 20vPnC | Cohort 3: 13vPnC
Started | 1514 | 1495 | 334 | 111 | 336 | 112
Evaluable 13-Matched Immunogenicity Population | 1435 | 1420 | 0 | 0 | 0 | 0
Evaluable 7-Additional Immunogenicity Population | 1433 | 1383 | 0 | 0 | 0 | 0
Vaccination 1 | 1507 | 1490 | 334 | 111 | 335 | 112
Vaccination 2 | 1461 | 1446 | 0 | 0 | 0 | 0
Safety Population | 1507 | 1490 | 334 | 111 | 335 | 112
Evaluable-20 Immunogenicity Population | 946 (Only for 60-64 years of age.) | 0 | 321 | 0 | 317 | 0
Completed | 1418 | 1417 | 323 | 109 | 319 | 104
Not Completed | 96 | 78 | 11 | 2 | 17 | 8
Not completed — Adverse Event | 11 | 8 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 41 | 28 | 9 | 2 | 14 | 8
Not completed — No longer met eligibility criteria | 3 | 9 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 21 | 13 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 19 | 20 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received 1 dose of any of the following: 20vPnC, 13vPnC, PPSV23 or saline and had safety follow-up after any vaccination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23 | Cohort 2: 20vPnC | Cohort 2: 13vPnC | Cohort 3: 20vPnC | Cohort 3: 13vPnC | Total
Number analyzed (Participants) | 1507 | 1490 | 334 | 111 | 335 | 112 | 3889
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (4.82) | 64.6 (4.81) | 54.9 (2.77) | 55.0 (3.11) | 34.0 (8.77) | 33.9 (8.03) | 60.0 (11.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 897 | 879 | 195 | 69 | 214 | 77 | 2331
  Male | 610 | 611 | 139 | 42 | 121 | 35 | 1558
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 167 | 169 | 12 | 8 | 24 | 7 | 387
  Not Hispanic or Latino | 1324 | 1308 | 319 | 101 | 300 | 102 | 3454
  Unknown or Not Reported | 16 | 13 | 3 | 2 | 11 | 3 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 9 | 0 | 3 | 1 | 1 | 20
  Asian | 19 | 15 | 10 | 2 | 11 | 1 | 58
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 3 | 1 | 6
  Black or African American | 177 | 212 | 35 | 15 | 34 | 7 | 480
  White | 1295 | 1237 | 278 | 90 | 274 | 101 | 3275
  More than one race | 7 | 9 | 6 | 1 | 8 | 1 | 32
  Unknown or Not Reported | 2 | 7 | 5 | 0 | 4 | 0 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 10 Days After Vaccination in All Cohorts
Description: Local reactions were recorded using an electronic diary. Local reactions included redness, swelling and pain at the injection site. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm). Redness and swelling were graded as mild (greater than [>] 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm) and severe (>10.0 cm). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), and severe (prevented daily activity).
Time Frame: Within 10 days after 20vPnC or 13vPnC
Population: Safety population included all participants who received 1 dose of any of the following: 20vPnC, 13vPnC, PPSV23 or saline and had safety follow-up after any vaccination. Here, "Overall Number of Participants Analyzed" =number of participants with any electronic diary data after 20vPnC or 13vPnC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23 | Cohort 2: 20vPnC | Cohort 2: 13vPnC | Cohort 3: 20vPnC | Cohort 3: 13vPnC
Number analyzed (Participants) | 1505 | 1483 | 331 | 111 | 335 | 112
percentage of participants
  Redness: Any | 7.3 [6.0 to 8.7] | 6.2 [5.0 to 7.6] | 8.2 [5.4 to 11.6] | 5.4 [2.0 to 11.4] | 9.0 [6.1 to 12.5] | 9.8 [5.0 to 16.9]
  Redness: Mild | 3.7 [2.8 to 4.8] | 3.8 [2.9 to 4.9] | 5.1 [3.0 to 8.1] | 2.7 [0.6 to 7.7] | 3.0 [1.4 to 5.4] | 5.4 [2.0 to 11.3]
  Redness: Moderate | 2.8 [2.0 to 3.8] | 2.2 [1.5 to 3.1] | 2.7 [1.3 to 5.1] | 2.7 [0.6 to 7.7] | 5.4 [3.2 to 8.4] | 4.5 [1.5 to 10.1]
  Redness: Severe | 0.8 [0.4 to 1.4] | 0.2 [0.0 to 0.6] | 0.3 [0.0 to 1.7] | 0 [0.0 to 3.3] | 0.6 [0.1 to 2.1] | 0 [0.0 to 3.2]
  Swelling: Any | 7.5 [6.2 to 9.0] | 8.0 [6.6 to 9.5] | 8.8 [5.9 to 12.3] | 10.8 [5.7 to 18.1] | 11.6 [8.4 to 15.6] | 12.5 [7.0 to 20.1]
  Swelling: Mild | 4.8 [3.8 to 6.0] | 4.9 [3.8 to 6.1] | 5.7 [3.5 to 8.8] | 7.2 [3.2 to 13.7] | 7.2 [4.6 to 10.5] | 8.9 [4.4 to 15.8]
  Swelling: Moderate | 2.4 [1.7 to 3.3] | 2.8 [2.0 to 3.8] | 3.0 [1.5 to 5.5] | 3.6 [1.0 to 9.0] | 4.5 [2.5 to 7.3] | 3.6 [1.0 to 8.9]
  Swelling: Severe | 0.3 [0.1 to 0.8] | 0.3 [0.1 to 0.7] | 0 [0.0 to 1.1] | 0 [0.0 to 3.3] | 0 [0.0 to 1.1] | 0 [0.0 to 3.2]
  Pain at the injection site: Any | 55.4 [52.9 to 57.9] | 54.1 [51.6 to 56.7] | 72.5 [67.4 to 77.2] | 69.4 [59.9 to 77.8] | 81.2 [76.6 to 85.2] | 82.1 [73.8 to 88.7]
  Pain at the injection site: Mild | 45.3 [42.8 to 47.9] | 44.6 [42.1 to 47.2] | 53.5 [47.9 to 58.9] | 52.3 [42.6 to 61.8] | 42.7 [37.3 to 48.2] | 52.7 [43.0 to 62.2]
  Pain at the injection site: Moderate | 9.9 [8.4 to 11.5] | 9.2 [7.7 to 10.8] | 17.8 [13.9 to 22.4] | 16.2 [9.9 to 24.4] | 38.2 [33.0 to 43.6] | 28.6 [20.4 to 37.9]
  Pain at the injection site: Severe | 0.2 [0.0 to 0.6] | 0.3 [0.1 to 0.8] | 1.2 [0.3 to 3.1] | 0.9 [0.0 to 4.9] | 0.3 [0.0 to 1.7] | 0.9 [0.0 to 4.9]

2. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination in All Cohorts
Description: Systemic events fever, fatigue, headache, muscle pain and joint pain were recorded by using an electronic diary. Fever was defined as greater than or equal to (>=) 38.0 degree Celsius (C) and categorized to >=38.0 to 38.4 degree C, >38.4 to 38.9 degree C, >38.9 to 40.0 degree C and >40.0 degree C. Fatigue, headache, muscle pain and joint pain were graded as mild (did not interfere with activity), moderate (some interference with activity) and severe (prevented daily routine activity).
Time Frame: Within 7 days after 20vPnC or 13vPnC
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23 | Cohort 2: 20vPnC | Cohort 2: 13vPnC | Cohort 3: 20vPnC | Cohort 3: 13vPnC
Number analyzed (Participants) | 1505 | 1483 | 331 | 111 | 335 | 112
percentage of participants
  Fever: >=38.0 degree C | 0.9 [0.5 to 1.6] | 0.8 [0.4 to 1.4] | 1.5 [0.5 to 3.5] | 0.9 [0.0 to 4.9] | 1.2 [0.3 to 3.0] | 1.8 [0.2 to 6.3]
  Fever: >=38.0 degree C to 38.4 degree C | 0.3 [0.1 to 0.7] | 0.4 [0.1 to 0.9] | 0.6 [0.1 to 2.2] | 0.9 [0.0 to 4.9] | 0.6 [0.1 to 2.1] | 0 [0.0 to 3.2]
  Fever: >38.4 degree C to 38.9 degree C | 0.3 [0.1 to 0.7] | 0.2 [0.0 to 0.6] | 0.3 [0.0 to 1.7] | 0 [0.0 to 3.3] | 0.3 [0.0 to 1.7] | 0 [0.0 to 3.2]
  Fever: >38.9 degree C to 40.0 degree C | 0.0 [0.0 to 0.4] | 0 [0.0 to 0.2] | 0.3 [0.0 to 1.7] | 0 [0.0 to 3.3] | 0.3 [0.0 to 1.7] | 1.8 [0.2 to 6.3]
  Fever: >40.0 degree C | 0.3 [0.1 to 0.8] | 0.2 [0.0 to 0.6] | 0.3 [0.0 to 1.7] | 0 [0.0 to 3.3] | 0 [0.0 to 1.1] | 0 [0.0 to 3.2]
  Fatigue: Any | 30.2 [27.9 to 32.6] | 30.7 [28.3 to 33.1] | 39.3 [34.0 to 44.8] | 36.0 [27.1 to 45.7] | 42.7 [37.3 to 48.2] | 43.8 [34.4 to 53.4]
  Fatigue: Mild | 16.1 [14.3 to 18.1] | 17.5 [15.6 to 19.6] | 21.1 [16.9 to 25.9] | 18.0 [11.4 to 26.4] | 18.8 [14.8 to 23.4] | 20.5 [13.5 to 29.2]
  Fatigue: Moderate | 12.8 [11.2 to 14.6] | 11.9 [10.3 to 13.7] | 17.2 [13.3 to 21.7] | 15.3 [9.2 to 23.4] | 22.1 [17.8 to 26.9] | 19.6 [12.7 to 28.2]
  Fatigue: Severe | 1.2 [0.7 to 1.9] | 1.2 [0.7 to 1.9] | 0.9 [0.2 to 2.6] | 2.7 [0.6 to 7.7] | 1.8 [0.7 to 3.9] | 3.6 [1.0 to 8.9]
  Headache: Any | 21.5 [19.5 to 23.7] | 23.3 [21.1 to 25.5] | 32.3 [27.3 to 37.7] | 36.0 [27.1 to 45.7] | 38.8 [33.6 to 44.3] | 33.9 [25.3 to 43.5]
  Headache: Mild | 15.5 [13.7 to 17.4] | 17.0 [15.1 to 19.0] | 20.5 [16.3 to 25.3] | 21.6 [14.4 to 30.4] | 21.5 [17.2 to 26.3] | 16.1 [9.8 to 24.2]
  Headache: Moderate | 5.4 [4.3 to 6.6] | 5.9 [4.8 to 7.3] | 10.9 [7.7 to 14.7] | 13.5 [7.8 to 21.3] | 14.6 [11.0 to 18.9] | 17.0 [10.5 to 25.2]
  Headache: Severe | 0.7 [0.3 to 1.2] | 0.3 [0.1 to 0.8] | 0.9 [0.2 to 2.6] | 0.9 [0.0 to 4.9] | 2.7 [1.2 to 5.0] | 0.9 [0.0 to 4.9]
  Muscle pain: Any | 39.1 [36.6 to 41.6] | 37.3 [34.8 to 39.8] | 49.8 [44.3 to 55.4] | 49.5 [39.9 to 59.2] | 66.6 [61.2 to 71.6] | 74.1 [65.0 to 81.9]
  Muscle pain: Mild | 28.9 [26.6 to 31.3] | 26.8 [24.6 to 29.2] | 33.8 [28.8 to 39.2] | 31.5 [23.0 to 41.0] | 36.4 [31.3 to 41.8] | 42.0 [32.7 to 51.7]
  Muscle pain: Moderate | 9.8 [8.3 to 11.4] | 10.0 [8.5 to 11.6] | 15.4 [11.7 to 19.8] | 17.1 [10.6 to 25.4] | 29.0 [24.2 to 34.1] | 31.3 [22.8 to 40.7]
  Muscle pain: Severe | 0.4 [0.1 to 0.9] | 0.5 [0.2 to 1.0] | 0.6 [0.1 to 2.2] | 0.9 [0.0 to 4.9] | 1.2 [0.3 to 3.0] | 0.9 [0.0 to 4.9]
  Joint pain: Any | 12.6 [11.0 to 14.4] | 13.7 [12.0 to 15.5] | 15.4 [11.7 to 19.8] | 20.7 [13.6 to 29.5] | 13.4 [10.0 to 17.6] | 17.9 [11.3 to 26.2]
  Joint pain: Mild | 6.9 [5.7 to 8.3] | 7.1 [5.9 to 8.6] | 10.6 [7.5 to 14.4] | 12.6 [7.1 to 20.3] | 6.3 [3.9 to 9.4] | 8.9 [4.4 to 15.8]
  Joint pain: Moderate | 5.4 [4.3 to 6.6] | 6.3 [5.2 to 7.7] | 4.8 [2.8 to 7.7] | 7.2 [3.2 to 13.7] | 7.2 [4.6 to 10.5] | 8.0 [3.7 to 14.7]
  Joint pain: Severe | 0.3 [0.1 to 0.8] | 0.2 [0.0 to 0.6] | 0 [0.0 to 1.1] | 0.9 [0.0 to 4.9] | 0 [0.0 to 1.1] | 0.9 [0.0 to 4.9]

3. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Vaccination in All Cohorts
Description: An AE was any untoward medical occurrence in study participants who received study vaccine without regard to possibility of causal relationship with the treatment.
Time Frame: Within 1 month after 20vPnC or 13vPnC
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23 | Cohort 2: 20vPnC | Cohort 2: 13vPnC | Cohort 3: 20vPnC | Cohort 3: 13vPnC
Number analyzed (Participants) | 1507 | 1490 | 334 | 111 | 335 | 112
percentage of participants | 9.8 [8.4 to 11.4] | 11.1 [9.6 to 12.8] | 10.2 [7.2 to 13.9] | 8.1 [3.8 to 14.8] | 15.2 [11.6 to 19.5] | 11.6 [6.3 to 19.0]

4. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Within 6 Months After Vaccination in All Cohorts
Description: An SAE was any untoward medical occurrence at any dose that results in death; is life-threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect or that is considered to be an important medical event.
Time Frame: Within 6 months after 20vPnC or 13vPnC
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23 | Cohort 2: 20vPnC | Cohort 2: 13vPnC | Cohort 3: 20vPnC | Cohort 3: 13vPnC
Number analyzed (Participants) | 1507 | 1490 | 334 | 111 | 335 | 112
percentage of participants | 2.4 [1.7 to 3.3] | 1.9 [1.3 to 2.8] | 0.3 [0.0 to 1.7] | 0.9 [0.0 to 4.9] | 0.6 [0.1 to 2.1] | 0.9 [0.0 to 4.9]

5. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Conditions (NDCMCs) Within 6 Months After Vaccination in All Cohorts
Description: An NDCMC was defined as a disease or medical condition, not previously identified, that was expected to be persistent or was otherwise long-lasting in its effects.
Time Frame: Within 6 months after 20vPnC or 13vPnC
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23 | Cohort 2: 20vPnC | Cohort 2: 13vPnC | Cohort 3: 20vPnC | Cohort 3: 13vPnC
Number analyzed (Participants) | 1507 | 1490 | 334 | 111 | 335 | 112
percentage of participants | 2.3 [1.6 to 3.1] | 2.3 [1.6 to 3.3] | 1.5 [0.5 to 3.5] | 0.9 [0.0 to 4.9] | 1.5 [0.5 to 3.4] | 1.8 [0.2 to 6.3]

6. Primary Outcome: Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for the 13 Matched Serotypes at 1 Month After Vaccination 1 (20vPnC or 13vPnC) in Cohort 1: Evaluable 13-Matched Immunogenicity Population
Description: OPA GMTs were determined for serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F. OPA titer was expressed as reciprocal of the highest serum dilution. OPA geometric mean and 2-sided 95% CIs were calculated.
Time Frame: 1 month after Vaccination 1
Population: Evaluable 13-matched immunogenicity population included participants who were enrolled in the appropriate cohort based on age, received Vaccination 1 as randomized, had at least 1 valid OPA titer for any of the 13 matched serotypes from the blood collection 27 to 49 days after Vaccination 1, had no other major protocol deviations. Number analyzed=participants evaluable for this outcome measure at specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23
Number analyzed (Participants) | 1435 | 1420
titer
  Serotype 1: number analyzed (Participants) | 1430 | 1419
  Serotype 1 | 123.4 [112.3 to 135.5] | 153.8 [140.2 to 168.8]
  Serotype 3: number analyzed (Participants) | 1415 | 1411
  Serotype 3 | 40.7 [38.0 to 43.6] | 47.8 [44.7 to 51.2]
  Serotype 4: number analyzed (Participants) | 1415 | 1409
  Serotype 4 | 508.7 [456.5 to 566.9] | 626.9 [563.5 to 697.4]
  Serotype 5: number analyzed (Participants) | 1418 | 1395
  Serotype 5 | 91.6 [83.4 to 100.5] | 109.7 [100.1 to 120.3]
  Serotype 6A: number analyzed (Participants) | 1403 | 1390
  Serotype 6A | 889.0 [795.0 to 994.1] | 1165.1 [1043.3 to 1301.0]
  Serotype 6B: number analyzed (Participants) | 1413 | 1401
  Serotype 6B | 1115.2 [1003.1 to 1239.8] | 1341.3 [1208.5 to 1488.8]
  Serotype 7F: number analyzed (Participants) | 1409 | 1391
  Serotype 7F | 968.8 [887.0 to 1058.3] | 1129.2 [1034.7 to 1232.4]
  Serotype 9V: number analyzed (Participants) | 1399 | 1391
  Serotype 9V | 1455.5 [1317.5 to 1608.0] | 1567.8 [1420.5 to 1730.5]
  Serotype 14: number analyzed (Participants) | 1418 | 1408
  Serotype 14 | 746.7 [679.0 to 821.2] | 746.7 [679.8 to 820.1]
  Serotype 18C: number analyzed (Participants) | 1420 | 1403
  Serotype 18C | 1252.6 [1123.1 to 1397.0] | 1482.3 [1330.5 to 1651.5]
  Serotype 19A: number analyzed (Participants) | 1420 | 1398
  Serotype 19A | 517.9 [472.2 to 568.0] | 645.3 [588.9 to 707.1]
  Serotype 19F: number analyzed (Participants) | 1421 | 1403
  Serotype 19F | 265.8 [240.2 to 294.1] | 333.3 [301.5 to 368.3]
  Serotype 23F: number analyzed (Participants) | 1424 | 1409
  Serotype 23F | 276.5 [242.5 to 315.2] | 335.1 [294.4 to 381.4]
Statistical Analysis 1: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 1: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — Noninferiority for a serotype was declared if the lower bound of the 2-sided 95% CI for the geometric mean ratio (GMR) for that serotype was greater than 0.5 (2-fold criterion); Ratio of GMTs = 0.80, 95% CI 2-sided [0.71 to 0.90]
Statistical Analysis 2: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 3: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — Noninferiority for a serotype was declared if the lower bound of the 2-sided 95% CI for the GMR for that serotype was greater than 0.5 (2-fold criterion); Ratio of GMTs = 0.85, 95% CI 2-sided [0.78 to 0.93]
Statistical Analysis 3: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 4: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.81, 95% CI 2-sided [0.71 to 0.93]
Statistical Analysis 4: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 5: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.83, 95% CI 2-sided [0.74 to 0.94]
Statistical Analysis 5: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 6A: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.76, 95% CI 2-sided [0.66 to 0.88]
Statistical Analysis 6: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 6B: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.83, 95% CI 2-sided [0.73 to 0.95]
Statistical Analysis 7: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 7F: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.86, 95% CI 2-sided [0.77 to 0.96]
Statistical Analysis 8: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 9V: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.93, 95% CI 2-sided [0.82 to 1.05]
Statistical Analysis 9: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 14: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.00, 95% CI 2-sided [0.89 to 1.13]
Statistical Analysis 10: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 18C: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.85, 95% CI 2-sided [0.74 to 0.97]
Statistical Analysis 11: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 19A: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.80, 95% CI 2-sided [0.71 to 0.90]
Statistical Analysis 12: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 19F: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.80, 95% CI 2-sided [0.70 to 0.91]
Statistical Analysis 13: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 23F: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.83, 95% CI 2-sided [0.70 to 0.97]

7. Primary Outcome: Pneumococcal OPA GMTs for the 7 Additional Serotypes at 1 Month After Vaccination 1 (20vPnC) or 1 Month After Vaccination 2 (PPSV23) in Cohort 1: Evaluable 7-Additional Immunogenicity Population (E7-AIP)
Description: OPA GMTs were determined for serotypes: 8, 10A, 11A, 12F, 15B, 22F and 33F. OPA titer was expressed as reciprocal of the highest serum dilution. OPA geometric mean and 2-sided 95% CIs were calculated.
Time Frame: 1 month after Vaccination 1 in "Cohort 1: 20vPnC/Saline"; 1 month after Vaccination 2 in "Cohort 1: 13vPnC/PPSV23"
Population: Evaluable 7-additional immunogenicity population: participants who were enrolled in the appropriate cohort based on age, received 20vPnC if randomized to 20vPnC/saline group or received both vaccinations if randomized to 13vPnC/PPSV23 group, had at least 1 valid OPA titers for any of the 7 additional serotypes from the blood collection 27 to 49 days after Vaccination 1 or Vaccination 2 respectively, had no other major protocol deviations. Number analyzed=participants evaluable at specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23
Number analyzed (Participants) | 1433 | 1383
titer
  Serotype 8: number analyzed (Participants) | 1374 | 1319
  Serotype 8 | 465.6 [422.5 to 513.1] | 848.1 [769.1 to 935.2]
  Serotype 10A: number analyzed (Participants) | 1310 | 1263
  Serotype 10A | 2007.6 [1808.0 to 2229.1] | 1079.9 [972.1 to 1199.7]
  Serotype 11A: number analyzed (Participants) | 1198 | 1209
  Serotype 11A | 4426.8 [3965.5 to 4941.8] | 2534.9 [2276.8 to 2822.3]
  Serotype 12F: number analyzed (Participants) | 1294 | 1222
  Serotype 12F | 2538.7 [2255.3 to 2857.7] | 1716.6 [1521.8 to 1936.3]
  Serotype 15B: number analyzed (Participants) | 1283 | 1249
  Serotype 15B | 2398.2 [2090.6 to 2751.2] | 768.5 [669.7 to 881.9]
  Serotype 22F: number analyzed (Participants) | 1274 | 1227
  Serotype 22F | 3666.2 [3244.4 to 4143.0] | 1846.2 [1636.6 to 2082.6]
  Serotype 33F: number analyzed (Participants) | 1157 | 1201
  Serotype 33F | 5125.9 [4611.3 to 5698.0] | 3720.6 [3356.2 to 4124.6]
Statistical Analysis 1: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 8: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.55, 95% CI 2-sided [0.49 to 0.62]
Statistical Analysis 2: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 10A: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.86, 95% CI 2-sided [1.63 to 2.12]
Statistical Analysis 3: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 11A: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.75, 95% CI 2-sided [1.52 to 2.01]
Statistical Analysis 4: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 12F: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.48, 95% CI 2-sided [1.27 to 1.72]
Statistical Analysis 5: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 15B: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 3.12, 95% CI 2-sided [2.62 to 3.71]
Statistical Analysis 6: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 22F: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.99, 95% CI 2-sided [1.70 to 2.32]
Statistical Analysis 7: Comparison: Cohort 1: 20vPnC/Saline vs Cohort 1: 13vPnC/PPSV23; Serotype 33F: Geometric mean ratio (20vPnC/Saline vs 13vPnC/PPSV23) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.38, 95% CI 2-sided [1.21 to 1.57]

8. Secondary Outcome: Pneumococcal OPA GMTs for the 20 Vaccines Serotypes at 1 Month After 20vPnC Vaccination in Cohort 2, 50 Through 59 Years of Age and Cohort 1, Only 60 Through 64 Years of Age: Evaluable-20 Immunogenicity Population
Description: OPA GMTs were determined for serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F and 33F. OPA titer was expressed as reciprocal of the highest serum dilution. OPA geometric mean and 2-sided 95% CIs were calculated.
Time Frame: 1 month after vaccination
Population: Evaluable-20 immunogenicity population included participants who were enrolled in the appropriate cohort based on age, received the vaccination as randomized, had at least 1 valid OPA titer from the blood collection 27 to 49 days after 20vPnC, had no other major protocol deviations. Number analyzed=participants evaluable at specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- Cohort 1: 20vPnC/Saline (60-64 Years of Age): Participants were randomized to receive a single dose of 0.5 milliliter (mL) intramuscular injection of 20-valent pneumococcal vaccine (20vPnC) at Vaccination 1 (Day 1) and a single dose of 0.5 mL intramuscular injection of saline at Vaccination 2 (28 to 42 days after Vaccination 1).
Arm/Group | Cohort 2: 20vPnC | Cohort 1: 20vPnC/Saline (60-64 Years of Age)
Number analyzed (Participants) | 321 | 946
titer
  Serotype 1: number analyzed (Participants) | 320 | 941
  Serotype 1 | 135.9 [113.1 to 163.4] | 131.8 [117.2 to 148.3]
  Serotype 3: number analyzed (Participants) | 318 | 935
  Serotype 3 | 43.3 [38.0 to 49.4] | 40.9 [37.6 to 44.5]
  Serotype 4: number analyzed (Participants) | 318 | 931
  Serotype 4 | 633.3 [513.9 to 780.4] | 577.9 [505.5 to 660.6]
  Serotype 5: number analyzed (Participants) | 313 | 935
  Serotype 5 | 84.6 [70.3 to 101.8] | 96.5 [85.8 to 108.6]
  Serotype 6A: number analyzed (Participants) | 318 | 921
  Serotype 6A | 1203.9 [968.1 to 1497.1] | 997.1 [866.5 to 1147.5]
  Serotype 6B: number analyzed (Participants) | 318 | 933
  Serotype 6B | 1502.7 [1228.2 to 1838.5] | 1199.0 [1054.3 to 1363.4]
  Serotype 7F: number analyzed (Participants) | 313 | 924
  Serotype 7F | 1047.0 [884.0 to 1240.2] | 1173.0 [1052.9 to 1306.9]
  Serotype 9V: number analyzed (Participants) | 312 | 922
  Serotype 9V | 1725.7 [1424.4 to 2090.6] | 1687.9 [1493.7 to 1907.3]
  Serotype 14: number analyzed (Participants) | 313 | 933
  Serotype 14 | 926.2 [761.8 to 1126.0] | 742.3 [655.8 to 840.2]
  Serotype 18C: number analyzed (Participants) | 315 | 937
  Serotype 18C | 1805.0 [1459.6 to 2232.2] | 1355.2 [1184.3 to 1550.7]
  Serotype 19A: number analyzed (Participants) | 318 | 932
  Serotype 19A | 618.4 [519.9 to 735.5] | 600.3 [537.5 to 670.6]
  Serotype 19F: number analyzed (Participants) | 320 | 937
  Serotype 19F | 286.7 [236.0 to 348.2] | 290.4 [256.4 to 329.0]
  Serotype 23F: number analyzed (Participants) | 319 | 937
  Serotype 23F | 549.1 [425.4 to 708.9] | 327.5 [278.2 to 385.6]
  Serotype 8: number analyzed (Participants) | 314 | 901
  Serotype 8 | 486.9 [400.6 to 591.9] | 502.3 [442.8 to 569.8]
  Serotype 10A: number analyzed (Participants) | 296 | 857
  Serotype 10A | 2520.4 [2076.0 to 3060.0] | 2437.0 [2149.8 to 2762.5]
  Serotype 11A: number analyzed (Participants) | 271 | 796
  Serotype 11A | 6416.9 [5131.9 to 8023.6] | 5248.9 [4564.5 to 6035.9]
  Serotype 12F: number analyzed (Participants) | 292 | 855
  Serotype 12F | 3445.1 [2807.8 to 4227.1] | 3105.2 [2722.7 to 3541.4]
  Serotype 15B: number analyzed (Participants) | 284 | 830
  Serotype 15B | 3355.9 [2582.0 to 4361.8] | 2873.7 [2438.1 to 3387.1]
  Serotype 22F: number analyzed (Participants) | 284 | 835
  Serotype 22F | 3808.1 [2998.2 to 4836.8] | 4228.4 [3629.6 to 4926.0]
  Serotype 33F: number analyzed (Participants) | 266 | 765
  Serotype 33F | 5571.3 [4495.7 to 6904.2] | 5445.2 [4749.2 to 6243.2]
Statistical Analysis 1: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 1: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.03, 95% CI 2-sided [0.84 to 1.26]
Statistical Analysis 2: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 3: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.06, 95% CI 2-sided [0.92 to 1.22]
Statistical Analysis 3: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 4: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.10, 95% CI 2-sided [0.87 to 1.38]
Statistical Analysis 4: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 5: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.88, 95% CI 2-sided [0.72 to 1.07]
Statistical Analysis 5: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 6A: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.21, 95% CI 2-sided [0.95 to 1.53]
Statistical Analysis 6: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 6B: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.25, 95% CI 2-sided [1.00 to 1.56]
Statistical Analysis 7: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 7F: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.89, 95% CI 2-sided [0.74 to 1.07]
Statistical Analysis 8: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 9V: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.02, 95% CI 2-sided [0.83 to 1.26]
Statistical Analysis 9: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 14: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.25, 95% CI 2-sided [1.01 to 1.54]
Statistical Analysis 10: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 18C: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.33, 95% CI 2-sided [1.06 to 1.68]
Statistical Analysis 11: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 19A: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.03, 95% CI 2-sided [0.85 to 1.25]
Statistical Analysis 12: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 19F: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.99, 95% CI 2-sided [0.80 to 1.22]
Statistical Analysis 13: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 23F: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.68, 95% CI 2-sided [1.27 to 2.22]
Statistical Analysis 14: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 8: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.97, 95% CI 2-sided [0.78 to 1.20]
Statistical Analysis 15: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 10A: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.03, 95% CI 2-sided [0.84 to 1.28]
Statistical Analysis 16: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 11A: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.22, 95% CI 2-sided [0.96 to 1.56]
Statistical Analysis 17: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 12F: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.11, 95% CI 2-sided [0.88 to 1.39]
Statistical Analysis 18: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 15B: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.17, 95% CI 2-sided [0.88 to 1.56]
Statistical Analysis 19: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 22F: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 0.90, 95% CI 2-sided [0.69 to 1.17]
Statistical Analysis 20: Comparison: Cohort 2: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 33F: GMR (20vPnC Cohort 2 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.02, 95% CI 2-sided [0.81 to 1.30]

9. Secondary Outcome: Pneumococcal OPA GMTs for the 20 Vaccines Serotypes at 1 Month After 20vPnC Vaccination in Cohort 3, 18 Through 49 Years and Cohort 1, Only 60 Through 64 Years of Age: Evaluable-20 Immunogenicity Population
Description: as for outcome 8
Time Frame: 1 month after vaccination
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 3: 20vPnC | Cohort 1: 20vPnC/Saline (60-64 Years of Age)
Number analyzed (Participants) | 317 | 946
titer
  Serotype 1: number analyzed (Participants) | 316 | 941
  Serotype 1 | 162.6 [135.1 to 195.6] | 132.0 [117.7 to 148.1]
  Serotype 3: number analyzed (Participants) | 316 | 935
  Serotype 3 | 42.1 [36.9 to 48.1] | 42.0 [38.7 to 45.7]
  Serotype 4: number analyzed (Participants) | 315 | 931
  Serotype 4 | 1966.7 [1599.5 to 2418.3] | 594.5 [522.9 to 675.9]
  Serotype 5: number analyzed (Participants) | 317 | 935
  Serotype 5 | 107.9 [89.4 to 130.1] | 96.9 [86.2 to 109.0]
  Serotype 6A: number analyzed (Participants) | 315 | 921
  Serotype 6A | 3930.5 [3176.0 to 4864.4] | 1022.8 [896.1 to 1167.4]
  Serotype 6B: number analyzed (Participants) | 314 | 933
  Serotype 6B | 4260.0 [3461.3 to 5243.1] | 1250.4 [1102.3 to 1418.4]
  Serotype 7F: number analyzed (Participants) | 311 | 924
  Serotype 7F | 1872.8 [1564.2 to 2242.4] | 1187.2 [1064.4 to 1324.2]
  Serotype 9V: number analyzed (Participants) | 315 | 922
  Serotype 9V | 6041.4 [4962.5 to 7354.9] | 1726.7 [1529.2 to 1949.7]
  Serotype 14: number analyzed (Participants) | 316 | 933
  Serotype 14 | 1848.4 [1514.7 to 2255.7] | 772.8 [684.7 to 872.3]
  Serotype 18C: number analyzed (Participants) | 312 | 937
  Serotype 18C | 4460.5 [3584.6 to 5550.4] | 1395.3 [1220.9 to 1594.5]
  Serotype 19A: number analyzed (Participants) | 312 | 932
  Serotype 19A | 1415.0 [1181.8 to 1694.2] | 611.3 [547.8 to 682.3]
  Serotype 19F: number analyzed (Participants) | 315 | 937
  Serotype 19F | 654.8 [538.2 to 796.8] | 301.2 [266.7 to 340.1]
  Serotype 23F: number analyzed (Participants) | 315 | 937
  Serotype 23F | 1559.2 [1208.1 to 2012.2] | 324.5 [277.1 to 380.1]
  Serotype 8: number analyzed (Participants) | 306 | 901
  Serotype 8 | 867.0 [709.7 to 1059.2] | 508.1 [448.8 to 575.3]
  Serotype 10A: number analyzed (Participants) | 292 | 857
  Serotype 10A | 4157.3 [3410.9 to 5067.0] | 2569.7 [2274.0 to 2903.7]
  Serotype 11A: number analyzed (Participants) | 263 | 796
  Serotype 11A | 7169.3 [5735.7 to 8961.1] | 5419.7 [4737.7 to 6199.7]
  Serotype 12F: number analyzed (Participants) | 273 | 855
  Serotype 12F | 5875.4 [4719.8 to 7314.1] | 3074.5 [2697.9 to 3503.7]
  Serotype 15B: number analyzed (Participants) | 279 | 830
  Serotype 15B | 4601.0 [3487.9 to 6069.4] | 3019.0 [2562.8 to 3556.4]
  Serotype 22F: number analyzed (Participants) | 273 | 835
  Serotype 22F | 7568.2 [5927.4 to 9663.2] | 4482.5 [3862.7 to 5201.8]
  Serotype 33F: number analyzed (Participants) | 251 | 765
  Serotype 33F | 7976.9 [6341.7 to 10033.7] | 5693.2 [4970.1 to 6521.5]
Statistical Analysis 1: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 1: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.23, 95% CI 2-sided [1.01 to 1.50]
Statistical Analysis 2: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 3: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.00, 95% CI 2-sided [0.87 to 1.16]
Statistical Analysis 3: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 4: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 3.31, 95% CI 2-sided [2.65 to 4.13]
Statistical Analysis 4: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 5: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.11, 95% CI 2-sided [0.91 to 1.36]
Statistical Analysis 5: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 6A: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 3.84, 95% CI 2-sided [3.06 to 4.83]
Statistical Analysis 6: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 6B: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 3.41, 95% CI 2-sided [2.73 to 4.26]
Statistical Analysis 7: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 7F: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.58, 95% CI 2-sided [1.30 to 1.91]
Statistical Analysis 8: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 9V: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 3.50, 95% CI 2-sided [2.83 to 4.33]
Statistical Analysis 9: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 14: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 2.39, 95% CI 2-sided [1.93 to 2.96]
Statistical Analysis 10: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 18C: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 3.20, 95% CI 2-sided [2.53 to 4.04]
Statistical Analysis 11: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 19A: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 2.31, 95% CI 2-sided [1.91 to 2.81]
Statistical Analysis 12: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 19F: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 2.17, 95% CI 2-sided [1.76 to 2.68]
Statistical Analysis 13: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 23F: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 4.80, 95% CI 2-sided [3.65 to 6.32]
Statistical Analysis 14: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 8: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.71, 95% CI 2-sided [1.38 to 2.12]
Statistical Analysis 15: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 10A: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.62, 95% CI 2-sided [1.31 to 2.00]
Statistical Analysis 16: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 11A: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.32, 95% CI 2-sided [1.04 to 1.68]
Statistical Analysis 17: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 12F: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.91, 95% CI 2-sided [1.51 to 2.41]
Statistical Analysis 18: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 15B: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.52, 95% CI 2-sided [1.13 to 2.05]
Statistical Analysis 19: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 22F: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.69, 95% CI 2-sided [1.30 to 2.20]
Statistical Analysis 20: Comparison: Cohort 3: 20vPnC vs Cohort 1: 20vPnC/Saline (60-64 Years of Age); Serotype 33F: GMR (20vPnC Cohort 3 vs 20vPnC Cohort 1 60-64 years of age) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; Ratio of GMTs = 1.40, 95% CI 2-sided [1.10 to 1.79]

10. Secondary Outcome: Pneumococcal OPA Geometric Mean Fold Rises (GMFRs) for the 13 Matched Serotypes From Before Vaccination 1 to 1 Month After Vaccination 1 (20vPnC or 13vPnC) in Cohort 1: Evaluable 13-Matched Immunogenicity Population
Description: OPA GMFR is the ratio of OPA GMT, 1 month after vaccination to before vaccination OPA GMT. OPA GMFRs from before to 1 month after vaccination were calculated along with corresponding 2-sided 95% CIs for pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F.
Time Frame: Before Vaccination 1 to 1 month after Vaccination 1
Population: Evaluable 13-matched immunogenicity population included participants who were enrolled in the appropriate cohort based on age, received Vaccination 1 as randomized, had at least 1 valid OPA titer for any of the 13 matched serotypes from the blood collection 27 to 49 days after Vaccination 1, had no other major protocol deviations. Number analyzed=participants evaluable with OPA titers available at both timepoints at the specified row.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23
Number analyzed (Participants) | 1435 | 1420
fold rise
  Serotype 1: number analyzed (Participants) | 1425 | 1418
  Serotype 1 | 12.6 [11.5 to 13.8] | 15.4 [14.1 to 16.8]
  Serotype 3: number analyzed (Participants) | 1404 | 1401
  Serotype 3 | 4.8 [4.5 to 5.2] | 5.8 [5.4 to 6.2]
  Serotype 4: number analyzed (Participants) | 1370 | 1374
  Serotype 4 | 31.2 [27.8 to 34.9] | 39.3 [35.1 to 44.1]
  Serotype 5: number analyzed (Participants) | 1411 | 1394
  Serotype 5 | 6.1 [5.6 to 6.6] | 7.2 [6.6 to 7.8]
  Serotype 6A: number analyzed (Participants) | 1382 | 1371
  Serotype 6A | 34.3 [30.7 to 38.3] | 42.6 [38.2 to 47.5]
  Serotype 6B: number analyzed (Participants) | 1360 | 1360
  Serotype 6B | 23.8 [21.3 to 26.6] | 26.5 [23.7 to 29.6]
  Serotype 7F: number analyzed (Participants) | 1367 | 1355
  Serotype 7F | 12.2 [11.1 to 13.3] | 13.5 [12.3 to 14.8]
  Serotype 9V: number analyzed (Participants) | 1317 | 1294
  Serotype 9V | 11.0 [9.9 to 12.2] | 12.5 [11.3 to 13.9]
  Serotype 14: number analyzed (Participants) | 1370 | 1366
  Serotype 14 | 9.3 [8.3 to 10.3] | 8.3 [7.4 to 9.2]
  Serotype 18C: number analyzed (Participants) | 1407 | 1396
  Serotype 18C | 33.8 [30.0 to 38.1] | 37.7 [33.5 to 42.5]
  Serotype 19A: number analyzed (Participants) | 1400 | 1379
  Serotype 19A | 21.0 [19.0 to 23.3] | 25.9 [23.3 to 28.8]
  Serotype 19F: number analyzed (Participants) | 1405 | 1397
  Serotype 19F | 8.6 [7.9 to 9.5] | 10.8 [9.8 to 11.9]
  Serotype 23F: number analyzed (Participants) | 1409 | 1402
  Serotype 23F | 24.9 [22.0 to 28.1] | 30.7 [27.1 to 34.7]

11. Secondary Outcome: Pneumococcal OPA GMFRs for the Additional 7 Serotypes From Before Vaccination 1 to 1 Month After Vaccination 1 (20vPnC) or From Before Vaccination 1 to 1 Month After Vaccination 2 (PPSV23) in Cohort 1: Evaluable 7-Additional Immunogenicity Population
Description: OPA GMFR is the ratio of OPA GMT, 1 month after vaccination to before vaccination OPA GMT. OPA GMFRs from before to 1 month after vaccination were calculated along with corresponding 2-sided 95% CIs for pneumococcal serotypes 8, 10A, 11A, 12F, 15B, 22F and 33F.
Time Frame: From before Vaccination 1 to 1 month after Vaccination 1 in "Cohort 1: 20vPnC/Saline" or From before Vaccination 1 to 1 month after Vaccination 2 in "Cohort 1: 13vPnC/PPSV23"
Population: E7-AIP included participants who were enrolled in appropriate cohort based on age, received 20vPnC if randomized to 20vPnC/saline group or received both vaccinations if randomized to 13vPnC/PPSV23 group, had at least 1 valid OPA titers for any of 7 additional serotypes from blood collection 27 to 49 days after Vaccination 1 or Vaccination 2 respectively, had no other major protocol deviations. Number analyzed=participants evaluable with OPA titers available at both timepoints at specified row.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23
Number analyzed (Participants) | 1433 | 1383
fold rise
  Serotype 8: number analyzed (Participants) | 1353 | 1293
  Serotype 8 | 22.1 [20.0 to 24.5] | 40.4 [36.6 to 44.7]
  Serotype 10A: number analyzed (Participants) | 1208 | 1164
  Serotype 10A | 18.5 [16.5 to 20.6] | 10.1 [9.1 to 11.3]
  Serotype 11A: number analyzed (Participants) | 973 | 993
  Serotype 11A | 9.3 [8.1 to 10.7] | 6.0 [5.3 to 6.9]
  Serotype 12F: number analyzed (Participants) | 1226 | 1147
  Serotype 12F | 72.4 [64.2 to 81.6] | 47.3 [41.4 to 54.1]
  Serotype 15B: number analyzed (Participants) | 1228 | 1178
  Serotype 15B | 55.4 [47.7 to 64.4] | 18.2 [15.6 to 21.1]
  Serotype 22F: number analyzed (Participants) | 1178 | 1156
  Serotype 22F | 78.5 [67.3 to 91.5] | 37.9 [32.7 to 43.9]
  Serotype 33F: number analyzed (Participants) | 1020 | 1080
  Serotype 33F | 7.5 [6.7 to 8.5] | 5.7 [5.1 to 6.3]

12. Secondary Outcome: Pneumococcal OPA GMFRs for the 20 Vaccines Serotypes From Before Vaccination to 1 Month After Vaccination in Cohort 2 and 3: Evaluable-20 Immunogenicity Population
Description: OPA GMFR is the ratio of OPA GMT, 1 month after vaccination to before vaccination OPA GMT. OPA GMFRs from before to 1 month after vaccination were calculated along with corresponding 2-sided 95% CIs for pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F and 33F.
Time Frame: Before vaccination to 1 month after vaccination
Population: Evaluable-20 immunogenicity population included participants who were enrolled in the appropriate cohort based on age, received the vaccination as randomized, had at least 1 valid OPA titer from the blood collection 27 to 49 days after 20vPnC, had no other major protocol deviations. Number analyzed=participants evaluable with OPA titers available at both timepoints at the specified row.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Cohort 2: 20vPnC | Cohort 3: 20vPnC
Number analyzed (Participants) | 321 | 317
fold rise
  Serotype 1: number analyzed (Participants) | 319 | 315
  Serotype 1 | 14.4 [12.0 to 17.3] | 18.6 [16.0 to 21.8]
  Serotype 3: number analyzed (Participants) | 317 | 312
  Serotype 3 | 5.1 [4.4 to 5.9] | 4.8 [4.2 to 5.5]
  Serotype 4: number analyzed (Participants) | 304 | 302
  Serotype 4 | 43.4 [34.4 to 54.9] | 131.8 [106.4 to 163.4]
  Serotype 5: number analyzed (Participants) | 312 | 315
  Serotype 5 | 5.9 [5.0 to 7.0] | 7.9 [6.7 to 9.4]
  Serotype 6A: number analyzed (Participants) | 312 | 305
  Serotype 6A | 50.3 [40.2 to 63.0] | 146.5 [120.6 to 178.0]
  Serotype 6B: number analyzed (Participants) | 299 | 286
  Serotype 6B | 31.7 [25.3 to 39.7] | 70.3 [55.7 to 88.7]
  Serotype 7F: number analyzed (Participants) | 300 | 284
  Serotype 7F | 12.8 [10.7 to 15.4] | 19.7 [16.1 to 24.3]
  Serotype 9V: number analyzed (Participants) | 288 | 281
  Serotype 9V | 12.1 [9.9 to 14.7] | 35.1 [27.9 to 44.2]
  Serotype 14: number analyzed (Participants) | 300 | 291
  Serotype 14 | 10.4 [8.3 to 13.0] | 14.6 [11.3 to 18.9]
  Serotype 18C: number analyzed (Participants) | 308 | 299
  Serotype 18C | 48.3 [37.9 to 61.5] | 111.8 [86.8 to 143.8]
  Serotype 19A: number analyzed (Participants) | 310 | 299
  Serotype 19A | 23.6 [19.2 to 29.1] | 39.1 [30.9 to 49.6]
  Serotype 19F: number analyzed (Participants) | 316 | 310
  Serotype 19F | 9.2 [7.6 to 11.3] | 17.8 [14.7 to 21.6]
  Serotype 23F: number analyzed (Participants) | 313 | 309
  Serotype 23F | 47.8 [37.2 to 61.3] | 118.2 [92.7 to 150.7]
  Serotype 8: number analyzed (Participants) | 310 | 300
  Serotype 8 | 23.9 [19.3 to 29.6] | 34.6 [27.8 to 43.0]
  Serotype 10A: number analyzed (Participants) | 273 | 260
  Serotype 10A | 17.9 [14.2 to 22.6] | 22.7 [17.8 to 29.0]
  Serotype 11A: number analyzed (Participants) | 213 | 220
  Serotype 11A | 10.4 [7.7 to 14.2] | 5.2 [3.9 to 6.9]
  Serotype 12F: number analyzed (Participants) | 279 | 252
  Serotype 12F | 107.3 [85.8 to 134.1] | 171.1 [135.1 to 216.8]
  Serotype 15B: number analyzed (Participants) | 263 | 248
  Serotype 15B | 72.1 [51.9 to 100.1] | 65.0 [44.8 to 94.4]
  Serotype 22F: number analyzed (Participants) | 256 | 241
  Serotype 22F | 63.5 [44.8 to 90.1] | 69.3 [48.4 to 99.4]
  Serotype 33F: number analyzed (Participants) | 233 | 213
  Serotype 33F | 9.1 [7.1 to 11.7] | 7.5 [5.8 to 9.7]

13. Secondary Outcome: Percentage of Participants With >=4-Fold Rise in Pneumococcal OPA Titers to the 13 Matched Serotypes From Before Vaccination 1 to 1 Month After Vaccination 1 (20vPnC or 13vPnC) in Cohort 1: Evaluable 13-Matched Immunogenicity Population
Description: Percentage of participants with a >=4-fold rise in serotype-specific pneumococcal OPA titers from before vaccination to 1 month after vaccination along with corresponding 2-sided 95% CIs were calculated for pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F.
Time Frame: Before Vaccination 1 to 1 month after Vaccination 1
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23
Number analyzed (Participants) | 1435 | 1420
percentage of participants
  Serotype 1: number analyzed (Participants) | 1425 | 1418
  Serotype 1 | 72.1 [69.7 to 74.4] | 74.8 [72.4 to 77.0]
  Serotype 3: number analyzed (Participants) | 1404 | 1401
  Serotype 3 | 56.1 [53.4 to 58.7] | 61.7 [59.1 to 64.2]
  Serotype 4: number analyzed (Participants) | 1370 | 1374
  Serotype 4 | 75.5 [73.2 to 77.8] | 79.6 [77.4 to 81.7]
  Serotype 5: number analyzed (Participants) | 1411 | 1394
  Serotype 5 | 55.6 [52.9 to 58.2] | 60.6 [58.0 to 63.2]
  Serotype 6A: number analyzed (Participants) | 1382 | 1371
  Serotype 6A | 80.5 [78.3 to 82.5] | 84.0 [82.0 to 85.9]
  Serotype 6B: number analyzed (Participants) | 1360 | 1360
  Serotype 6B | 75.7 [73.3 to 77.9] | 77.6 [75.3 to 79.8]
  Serotype 7F: number analyzed (Participants) | 1367 | 1355
  Serotype 7F | 71.8 [69.3 to 74.1] | 72.3 [69.8 to 74.6]
  Serotype 9V: number analyzed (Participants) | 1317 | 1294
  Serotype 9V | 67.7 [65.1 to 70.3] | 69.3 [66.7 to 71.8]
  Serotype 14: number analyzed (Participants) | 1370 | 1366
  Serotype 14 | 58.2 [55.5 to 60.8] | 54.0 [51.3 to 56.6]
  Serotype 18C: number analyzed (Participants) | 1407 | 1396
  Serotype 18C | 77.7 [75.4 to 79.8] | 79.6 [77.4 to 81.7]
  Serotype 19A: number analyzed (Participants) | 1400 | 1379
  Serotype 19A | 73.6 [71.3 to 75.9] | 77.5 [75.2 to 79.7]
  Serotype 19F: number analyzed (Participants) | 1405 | 1397
  Serotype 19F | 63.6 [61.1 to 66.2] | 66.9 [64.4 to 69.4]
  Serotype 23F: number analyzed (Participants) | 1409 | 1402
  Serotype 23F | 70.6 [68.2 to 73.0] | 74.4 [72.0 to 76.7]

14. Secondary Outcome: Percentage of Participants With >=4-Fold Rise in Pneumococcal OPA Titers for the 7 Additional Serotypes From Before Vaccination 1 to 1 Month After Vaccination 1(20vPnC) or From Before Vaccination 1 to 1 Month After Vaccination 2(PPSV23) in Cohort 1:E7-AIP
Description: Percentage of participants with a >=4-fold rise in serotype-specific pneumococcal OPA titers from before vaccination to 1 month after vaccination along with corresponding 2-sided 95% CIs were calculated for pneumococcal serotypes 8, 10A, 11A, 12F, 15B, 22F and 33F.
Time Frame: Before Vaccination 1 to 1 month after Vaccination 1 for "Cohort 1: 20vPnC/Saline"; Before Vaccination 1 to 1 month after Vaccination 2 for "Cohort 1: 13vPnC/PPSV23"
Population: E7-AIP included participants who were enrolled in appropriate cohort based on age, received 20vPnC if randomized to 20vPnC/saline group or received both vaccinations if randomized to 13vPnC/PPSV23 group, had at least 1 valid OPA titers for any of 7 additional serotypes from blood collection 27 to 49 days after Vaccination 1 or Vaccination 2 respectively, had no other major protocol deviations. Number analyzed= participants evaluable at specified rows.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23
Number analyzed (Participants) | 1433 | 1383
percentage of participants
  Serotype 8: number analyzed (Participants) | 1353 | 1293
  Serotype 8 | 77.8 [75.5 to 80.0] | 86.8 [84.8 to 88.6]
  Serotype 10A: number analyzed (Participants) | 1208 | 1164
  Serotype 10A | 75.5 [73.0 to 77.9] | 65.6 [62.8 to 68.4]
  Serotype 11A: number analyzed (Participants) | 973 | 993
  Serotype 11A | 59.2 [56.0 to 62.3] | 51.9 [48.7 to 55.0]
  Serotype 12F: number analyzed (Participants) | 1226 | 1147
  Serotype 12F | 87.4 [85.5 to 89.2] | 80.6 [78.1 to 82.8]
  Serotype 15B: number analyzed (Participants) | 1228 | 1178
  Serotype 15B | 77.8 [75.3 to 80.1] | 63.8 [61.0 to 66.6]
  Serotype 22F: number analyzed (Participants) | 1178 | 1156
  Serotype 22F | 82.7 [80.4 to 84.8] | 76.8 [74.3 to 79.2]
  Serotype 33F: number analyzed (Participants) | 1020 | 1080
  Serotype 33F | 60.1 [57.0 to 63.1] | 55.5 [52.4 to 58.5]

15. Secondary Outcome: Percentage of Participants With >=4-Fold Rise in Pneumococcal OPA Titers for the 20 Vaccines Serotypes From Before Vaccination to 1 Month After Vaccination in Cohort 2 and 3: Evaluable-20 Immunogenicity Population
Description: Percentage of participants with a >=4-fold rise in serotype-specific pneumococcal OPA titers from before vaccination to 1 month after vaccination along with corresponding 2-sided 95% CIs were calculated for pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F and 33F.
Time Frame: Before vaccination to 1 month after vaccination
Population: Evaluable-20 immunogenicity population included participants who were enrolled in the appropriate cohort based on age, received the vaccination as randomized, had at least 1 valid OPA titer from the blood collection 27 to 49 days after 20vPnC, had no other major protocol deviations. Number analyzed =participants evaluable at specified rows.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: 20vPnC | Cohort 3: 20vPnC
Number analyzed (Participants) | 321 | 317
percentage of participants
  Serotype 1: number analyzed (Participants) | 319 | 315
  Serotype 1 | 74.9 [69.8 to 79.6] | 86.0 [81.7 to 89.7]
  Serotype 3: number analyzed (Participants) | 317 | 312
  Serotype 3 | 59.0 [53.4 to 64.5] | 56.7 [51.0 to 62.3]
  Serotype 4: number analyzed (Participants) | 304 | 302
  Serotype 4 | 84.2 [79.6 to 88.1] | 91.4 [87.6 to 94.3]
  Serotype 5: number analyzed (Participants) | 312 | 315
  Serotype 5 | 54.8 [49.1 to 60.4] | 64.8 [59.2 to 70.0]
  Serotype 6A: number analyzed (Participants) | 312 | 305
  Serotype 6A | 85.9 [81.5 to 89.6] | 96.7 [94.1 to 98.4]
  Serotype 6B: number analyzed (Participants) | 299 | 286
  Serotype 6B | 78.9 [73.9 to 83.4] | 89.2 [85.0 to 92.5]
  Serotype 7F: number analyzed (Participants) | 300 | 284
  Serotype 7F | 73.0 [67.6 to 77.9] | 76.1 [70.7 to 80.9]
  Serotype 9V: number analyzed (Participants) | 288 | 281
  Serotype 9V | 73.6 [68.1 to 78.6] | 84.0 [79.2 to 88.1]
  Serotype 14: number analyzed (Participants) | 300 | 291
  Serotype 14 | 62.3 [56.6 to 67.8] | 62.2 [56.4 to 67.8]
  Serotype 18C: number analyzed (Participants) | 308 | 299
  Serotype 18C | 82.5 [77.8 to 86.5] | 87.3 [83.0 to 90.8]
  Serotype 19A: number analyzed (Participants) | 310 | 299
  Serotype 19A | 80.0 [75.1 to 84.3] | 82.6 [77.8 to 86.7]
  Serotype 19F: number analyzed (Participants) | 316 | 310
  Serotype 19F | 64.2 [58.7 to 69.5] | 78.4 [73.4 to 82.8]
  Serotype 23F: number analyzed (Participants) | 313 | 309
  Serotype 23F | 81.2 [76.4 to 85.3] | 87.7 [83.5 to 91.1]
  Serotype 8: number analyzed (Participants) | 310 | 300
  Serotype 8 | 79.4 [74.4 to 83.7] | 83.0 [78.3 to 87.1]
  Serotype 10A: number analyzed (Participants) | 273 | 260
  Serotype 10A | 78.8 [73.4 to 83.5] | 78.8 [73.4 to 83.6]
  Serotype 11A: number analyzed (Participants) | 213 | 220
  Serotype 11A | 61.0 [54.1 to 67.6] | 47.3 [40.5 to 54.1]
  Serotype 12F: number analyzed (Participants) | 279 | 252
  Serotype 12F | 93.2 [89.6 to 95.9] | 93.7 [89.9 to 96.3]
  Serotype 15B: number analyzed (Participants) | 263 | 248
  Serotype 15B | 82.5 [77.4 to 86.9] | 73.4 [67.4 to 78.8]
  Serotype 22 F: number analyzed (Participants) | 256 | 241
  Serotype 22 F | 80.5 [75.1 to 85.1] | 83.8 [78.5 to 88.2]
  Serotype 33F: number analyzed (Participants) | 233 | 213
  Serotype 33F | 63.9 [57.4 to 70.1] | 60.6 [53.7 to 67.2]

16. Secondary Outcome: Percentage of Participants With Pneumococcal OPA Titers >= Lower Limit of Quantitation (LLOQ) for the 13 Matched Serotypes at 1 Month After Vaccination 1 (20vPnC or 13vPnC) in Cohort 1: Evaluable 13-Matched Immunogenicity Population
Description: The percentage of participants with OPA titers >=LLOQ along with corresponding 2-sided 95% CIs were calculated 1 month after vaccination for pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F.
Time Frame: 1 month after Vaccination 1
Population: Evaluable 13-matched immunogenicity population included participants who were enrolled in the appropriate cohort based on age, received Vaccination 1 as randomized, had at least 1 valid OPA titer for any of the 13 matched serotypes from the blood collection 27 to 49 days after Vaccination 1, had no other major protocol deviations. Number analyzed =participants evaluable for this outcome measure at specified rows.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23
Number analyzed (Participants) | 1435 | 1420
percentage of participants
  Serotype 1: number analyzed (Participants) | 1430 | 1419
  Serotype 1 | 85.0 [83.0 to 86.8] | 87.9 [86.1 to 89.5]
  Serotype 3: number analyzed (Participants) | 1415 | 1411
  Serotype 3 | 84.2 [82.2 to 86.0] | 87.0 [85.2 to 88.7]
  Serotype 4: number analyzed (Participants) | 1415 | 1409
  Serotype 4 | 91.1 [89.5 to 92.5] | 92.1 [90.5 to 93.4]
  Serotype 5: number analyzed (Participants) | 1418 | 1395
  Serotype 5 | 71.9 [69.5 to 74.3] | 76.0 [73.7 to 78.2]
  Serotype 6A: number analyzed (Participants) | 1403 | 1390
  Serotype 6A | 88.9 [87.1 to 90.5] | 90.9 [89.2 to 92.3]
  Serotype 6B: number analyzed (Participants) | 1413 | 1401
  Serotype 6B | 90.5 [88.9 to 92.0] | 91.6 [90.0 to 93.0]
  Serotype 7F: number analyzed (Participants) | 1409 | 1391
  Serotype 7F | 89.1 [87.3 to 90.7] | 91.3 [89.7 to 92.7]
  Serotype 9V: number analyzed (Participants) | 1399 | 1391
  Serotype 9V | 89.1 [87.4 to 90.7] | 90.3 [88.6 to 91.8]
  Serotype 14: number analyzed (Participants) | 1418 | 1408
  Serotype 14 | 91.6 [90.0 to 93.0] | 93.5 [92.1 to 94.8]
  Serotype 18C: number analyzed (Participants) | 1420 | 1403
  Serotype 18C | 93.8 [92.4 to 95.0] | 94.7 [93.4 to 95.8]
  Serotype 19A: number analyzed (Participants) | 1420 | 1398
  Serotype 19A | 96.3 [95.2 to 97.3] | 96.6 [95.5 to 97.5]
  Serotype 19F: number analyzed (Participants) | 1421 | 1403
  Serotype 19F | 80.3 [78.1 to 82.3] | 81.5 [79.3 to 83.5]
  Serotype 23F: number analyzed (Participants) | 1424 | 1409
  Serotype 23F | 82.1 [80.0 to 84.1] | 83.7 [81.6 to 85.6]

17. Secondary Outcome: Percentage of Participants With Pneumococcal OPA Titers >=LLOQ for the 7 Additional Serotypes at 1 Month After Vaccination 1 (20vPnC) or 1 Month After Vaccination 2 (PPSV23) in Cohort 1: Evaluable 7-Additional Immunogenicity Population
Description: The percentage of participants with OPA titers >=LLOQ along with corresponding 2-sided 95% CIs were calculated 1 month after vaccination for pneumococcal serotypes 8, 10A, 11A, 12F, 15B, 22F and 33F.
Time Frame: 1 month after Vaccination 1 in "Cohort 1: 20vPnC/Saline" or 1 month after Vaccination 2 in "Cohort 1: 13vPnC/PPSV23"
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23
Number analyzed (Participants) | 1433 | 1383
percentage of participants
  Serotype 8: number analyzed (Participants) | 1374 | 1319
  Serotype 8 | 92.9 [91.5 to 94.2] | 96.6 [95.5 to 97.5]
  Serotype 10A: number analyzed (Participants) | 1310 | 1263
  Serotype 10A | 95.6 [94.3 to 96.6] | 88.9 [87.1 to 90.6]
  Serotype 11A: number analyzed (Participants) | 1198 | 1209
  Serotype 11A | 97.7 [96.6 to 98.4] | 95.4 [94.0 to 96.5]
  Serotype 12F: number analyzed (Participants) | 1294 | 1222
  Serotype 12F | 95.7 [94.4 to 96.7] | 89.3 [87.4 to 91.0]
  Serotype 15B: number analyzed (Participants) | 1283 | 1249
  Serotype 15B | 94.1 [92.6 to 95.3] | 83.3 [81.1 to 85.3]
  Serotype 22F: number analyzed (Participants) | 1274 | 1227
  Serotype 22F | 98.6 [97.8 to 99.2] | 94.5 [93.0 to 95.7]
  Serotype 33F: number analyzed (Participants) | 1157 | 1201
  Serotype 33F | 96.4 [95.1 to 97.4] | 92.8 [91.2 to 94.2]

18. Secondary Outcome: Percentage of Participants With Pneumococcal OPA Titers >=LLOQ for the 20 Vaccines Serotypes at 1 Month After Vaccination (20vPnC) in Cohort 2 and 3: Evaluable-20 Immunogenicity Population
Description: The percentage of participants with OPA titers >=LLOQ along with corresponding 2-sided 95% CIs were calculated 1 month after vaccination for pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 8, 10A, 11A, 12F, 15B, 22F and 33F. Data for this outcome measure were planned to be analyzed for the 20vPnC groups of Cohorts 2 and 3 only.
Time Frame: 1 month after vaccination
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: 20vPnC | Cohort 3: 20vPnC
Number analyzed (Participants) | 321 | 317
percentage of participants
  Serotype 1: number analyzed (Participants) | 320 | 316
  Serotype 1 | 87.2 [83.0 to 90.6] | 92.1 [88.5 to 94.8]
  Serotype 3: number analyzed (Participants) | 318 | 316
  Serotype 3 | 87.4 [83.3 to 90.9] | 89.9 [86.0 to 93.0]
  Serotype 4: number analyzed (Participants) | 318 | 315
  Serotype 4 | 94.0 [90.8 to 96.4] | 98.1 [95.9 to 99.3]
  Serotype 5: number analyzed (Participants) | 313 | 317
  Serotype 5 | 72.8 [67.6 to 77.7] | 81.1 [76.3 to 85.2]
  Serotype 6A: number analyzed (Participants) | 318 | 315
  Serotype 6A | 91.8 [88.2 to 94.6] | 99.7 [98.2 to 100.0]
  Serotype 6B: number analyzed (Participants) | 318 | 314
  Serotype 6B | 95.3 [92.3 to 97.3] | 99.0 [97.2 to 99.8]
  Serotype 7F: number analyzed (Participants) | 313 | 311
  Serotype 7F | 92.7 [89.2 to 95.3] | 93.9 [90.6 to 96.3]
  Serotype 9V: number analyzed (Participants) | 312 | 315
  Serotype 9V | 92.6 [89.1 to 95.3] | 99.0 [97.2 to 99.8]
  Serotype 14: number analyzed (Participants) | 313 | 316
  Serotype 14 | 94.9 [91.8 to 97.1] | 99.1 [97.3 to 99.8]
  Serotype 18C: number analyzed (Participants) | 315 | 312
  Serotype 18C | 97.5 [95.1 to 98.9] | 98.1 [95.9 to 99.3]
  Serotype 19A: number analyzed (Participants) | 318 | 312
  Serotype 19A | 98.7 [96.8 to 99.7] | 99.7 [98.2 to 100.0]
  Serotype 19F: number analyzed (Participants) | 320 | 315
  Serotype 19F | 81.9 [77.2 to 85.9] | 95.2 [92.3 to 97.3]
  Serotype 23F: number analyzed (Participants) | 319 | 315
  Serotype 23F | 89.3 [85.4 to 92.5] | 96.5 [93.8 to 98.2]
  Serotype 8: number analyzed (Participants) | 314 | 306
  Serotype 8 | 92.4 [88.8 to 95.0] | 95.8 [92.8 to 97.7]
  Serotype 10A: number analyzed (Participants) | 296 | 292
  Serotype 10A | 98.3 [96.1 to 99.4] | 100.0 [98.7 to 100.0]
  Serotype 11A: number analyzed (Participants) | 271 | 263
  Serotype 11A | 97.0 [94.3 to 98.7] | 99.6 [97.9 to 100.0]
  Serotype 12F: number analyzed (Participants) | 292 | 273
  Serotype 12F | 97.9 [95.6 to 99.2] | 98.5 [96.3 to 99.6]
  Serotype 15B: number analyzed (Participants) | 284 | 279
  Serotype 15B | 95.8 [92.7 to 97.8] | 96.8 [94.0 to 98.5]
  Serotype 22F: number analyzed (Participants) | 284 | 273
  Serotype 22F | 98.2 [95.9 to 99.4] | 99.6 [98.0 to 100.0]
  Serotype 33F: number analyzed (Participants) | 266 | 251
  Serotype 33F | 95.9 [92.7 to 97.9] | 99.6 [97.8 to 100.0]

ADVERSE EVENTS:
Time Frame: Local reactions: within 10 days after Vaccination 1 (systematic assessment), Systemic events: within 7 days after Vaccination 1 (systematic assessment), Non serious AEs: up to 1 month after Vaccination 1, SAEs: up to 6 months after Vaccination 1
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety population was used for the analysis.
Arm/Group | Cohort 1: 20vPnC/Saline | Cohort 1: 13vPnC/PPSV23 | Cohort 2: 20vPnC | Cohort 2: 13vPnC | Cohort 3: 20vPnC | Cohort 3: 13vPnC
All-Cause Mortality (participants affected / at risk) | 1/1507 | 0/1490 | 0/334 | 0/111 | 0/335 | 0/112
Serious Adverse Events (participants affected / at risk) | 36/1507 | 29/1490 | 1/334 | 1/111 | 2/335 | 1/112
Other Adverse Events (participants affected / at risk) | 1074/1507 | 1063/1490 | 281/334 | 91/111 | 302/335 | 107/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 20vPnC/Saline (N=1507) | Cohort 1: 13vPnC/PPSV23 (N=1490) | Cohort 2: 20vPnC (N=334) | Cohort 2: 13vPnC (N=111) | Cohort 3: 20vPnC (N=335) | Cohort 3: 13vPnC (N=112)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 3 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Silent myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Biloma (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Device malfunction (Product Issues) | 0 | 1 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0
End stage renal disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Herpes simplex meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 20vPnC/Saline (N=1507) | Cohort 1: 13vPnC/PPSV23 (N=1490) | Cohort 2: 20vPnC (N=334) | Cohort 2: 13vPnC (N=111) | Cohort 3: 20vPnC (N=335) | Cohort 3: 13vPnC (N=112)
Fatigue (FATIGUE) (General disorders) | 454 | 455 | 130 | 40 | 143 | 49
Injection site erythema (REDNESS) (General disorders) | 110 | 92 | 27 | 6 | 30 | 11
Injection site pain (PAIN) (General disorders) | 834 | 803 | 240 | 77 | 272 | 92
Injection site swelling (SWELLING) (General disorders) | 113 | 118 | 29 | 12 | 39 | 14
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 190 | 203 | 51 | 23 | 45 | 20
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 588 | 553 | 165 | 55 | 223 | 83
Headache (HEADACHE) (Nervous system disorders) | 324 | 345 | 107 | 40 | 130 | 38
Pyrexia (FEVER) (General disorders) | 0 | 0 | 5 | 1 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 4 | 3 | 7 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 7 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 6 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT03760146/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT03760146/SAP_001.pdf